CLINICAL TRIAL: NCT05554380
Title: Phase 2 Study of Paclitaxel (NSC #673089) + Ipatasertib (NSC #781451) in Taxane-Refractory Participants With PTEN/AKT-Altered Advanced Non-Breast Solid Tumors: A ComboMATCH Treatment Trial
Brief Title: Study of Chemotherapy Plus Ipatasertib for People With Solid Tumors With PTEN/AKT Mutations, A ComboMATCH Treatment Trial
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - study has reached accrual goal for analysis
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07304; NCI-2022-07304 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-S3 (Other: SWOG); EAY191-S3 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; ipatasertib; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (paclitaxel, ipatasertib) (Experimental): Patients receive paclitaxel IV on days 1, 8, and 15 and ipatasertib PO on days 1-21 of each cycle. Treatment repeats every 28 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a CT or MRI and blood collection throughout the trial. Patients also undergo a tumor biopsy during screening and optionally during follow-up.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II ComboMATCH treatment trial tests the usual treatment of chemotherapy (paclitaxel) plus ipatasertib in patients with solid tumor cancers that that cannot be removed by surgery (unresectable), has spread to nearby tissue or lymph nodes (locally advanced) or from where it first started (primary site) to other places in the body (metastatic), and has PTEN and AKT genetic changes. Chemotherapy drugs, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Targeted therapy, such as Ipatasertib, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The addition of ipatasertib to paclitaxel in solid tumors with PTEN and AKT genetic changes could increase the percentage of tumors that shrink as well as lengthen the time that the tumors remain stable (without progression). Researchers hope to learn if paclitaxel plus ipatasertib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the overall response rate (ORR) (confirmed and unconfirmed, complete, and partial) with the combination of paclitaxel plus ipatasertib in participants with advanced PTEN/AKT-altered non-breast solid tumors who have previously progressed on taxane-based therapy

SECONDARY OBJECTIVES:

I. To assess the progression-free survival (PFS) in the study population. II. To assess the duration of response (DoR) in participants who respond to treatment.

III. To assess the overall survival (OS) in the study population. IV. To evaluate the frequency and severity of toxicities related to the combination therapy.

V. Collect tissue and provide it to the ComboMATCH Registration protocol to assess concordance between the diagnostic tumor mutation profile generated by the designated laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration protocol. For this treatment substudy, the outcome objective will be to report the proportion of cases providing sufficient tissue for that integrated scientific activity in the ComboMATCH Registration protocol.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To conduct whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing (RNAseq) analysis of tumors at baseline (mandatory), as well as PTEN expression analysis of tumors at baseline (2nd priority after nucleic acid for WES and RNAseq).

II. To explore changes in plasma PTEN/AKT mutation allelic burden and other molecular findings at baseline (mandatory) and upon progression (optional) using ctDNA and correlate changes with response/resistance to therapy.

III. To perform comprehensive protein expression and function analysis on fresh frozen specimens (optional) collected at baseline and at progression to assess determinants of response and resistance to therapy.

OUTLINE:

Patients receive paclitaxel intravenously (IV) on days 1, 8, and 15 and ipatasertib orally (PO) on days 1-21 of each cycle. Treatment repeats every 28 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo a computed tomography (CT) or magnetic resonance imaging (MRI) and blood collection throughout the trial. Patients also undergo a tumor biopsy during screening and optionally during follow-up.

After completion of study treatment, patients are followed until death or 3 years after registration, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-S3 based on the presence of an actionable mutation as defined in EAY191
* GENERAL COMBOMATCH EAY191 REGISTRATION INCLUSION CRITERIA:
* Participants must be enrolled on the ComboMATCH Master Registration Trial EAY191
* Participants must have an activating AKT mutation (a known mutation in AKT1, AKT2, or AKT3, a single nucleotide variant, insertion, or deletion), PTEN mutation (a known mutation in PTEN, a single nucleotide variant, insertion, or deletion), or genomic deletion loss of PTEN as determined by the ComboMATCH screening assessment
* GENERAL COMBOMATCH EAY191 REGISTRATION EXCLUSION CRITERIA:
* Participants must not have an activating KRAS, NRAS, HRAS, or BRAF mutation (a single nucleotide variant, insertion, or deletion) as determined by the ComboMATCH screening assessment
* Participants must have disease that can be safely biopsied and agree to a pre-treatment biopsy or have archival tissue available from within 12 months prior to the date of registration on the ComboMATCH Registration Trial (EAY191)
* Participants must have a histologically confirmed non-breast solid malignancy
* Participants must have locally advanced, unresectable, or metastatic disease in the opinion of the treating investigator
* Participants must have measurable disease documented by CT or MRI. Measurable disease must be assessed within 28 days prior to registration. Non-measurable disease must be assessed within 42 days prior to registration. The CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1). Participants whose only measurable disease is within a previous radiation therapy port must demonstrate clearly progressive disease (in the opinion of the treating investigator) prior to registration
* Participants with known brain metastases must have a CT/MRI scan to evaluate for central nervous system (CNS) disease and show no evidence of progression within 42 days prior to registration
* Participants must have completed any CNS-directed therapy and/or local therapy for spinal cord compression at least 28 days prior to registration
* Participants must not have spinal cord compression or brain metastases unless: (1) metastases have been locally treated and have remained clinically controlled and asymptomatic for at least 14 days prior to registration, AND (2) participant has no residual neurological dysfunction and has been off corticosteroids for at least 24 hours prior to registration
* Participants must not have leptomeningeal disease
* Participants must have progressed on or within 6 months of taxane-based therapy in the neoadjuvant/adjuvant or metastatic setting prior to registration
* Participants must not have received any prior AKT inhibitor (e.g., capivasertib or ipatasertib); prior PI3K/mTOR inhibitor is acceptable
* Participants must not have received cancer-directed therapy prior for at least 14 days prior to initiation of treatment on study
* Participants must not be planning to receive any concurrent chemotherapy, immunotherapy, biologic, radiation, or hormonal therapy for cancer treatment while receiving treatment on this study
* Participants must be >= 18 years of age
* Participants must be able to swallow oral medications whole
* Participants must have a pre-study history and physical exam done within 28 days prior to registration
* Participants must have a Zubrod performance status of 0-2 within 28 days prior to registration
* Participants must have adverse events resolved =< grade 1 related to any prior therapy, except alopecia within 14 days prior to registration
* Participants with neuropathy must have resolved to < grade 2 within 14 days prior to registration
* Leukocytes >= 3 x 10^3/uL (within 28 days prior to registration)
* Absolute neutrophil count >= 1.5 x 10^3/uL (within 28 days prior to registration)
* Platelets >= 100 x 10^3/uL (within 28 days prior to registration)
* Total bilirubin =< institutional upper limit of normal (ULN) unless history of Gilbert's disease. Participants with history of Gilbert's disease must have total bilirubin =< 5 x institutional ULN (within 28 days prior to registration)
* Aspartate aminotransferase (AST) & alanine aminotransferase (ALT) =< 3 x institutional ULN (within 28 days prior to registration)
* Participants must have adequate cardiac function, class IIB (2B) or better. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification
* Participants must have a measured OR calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault formula. This specimen must have been drawn within 28 days prior to registration
* Participants with known human immunodeficiency virus (HIV)-infection must be receiving anti-retroviral therapy and have an undetectable viral load test on the most recent test results obtained within 6 months prior to registration
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within 28 days prior to registration
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to registration
* Participants must have an electrocardiography (ECG) performed (if clinically indicated with a corrected QTc interval of =< 470 msec) within 28 days prior to registration
* Participants must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ipatasertib and/or paclitaxel
* Participants must not have an active small/large bowel inflammation such as ulcerative colitis or Crohn's disease
* Participants must not have grade 2 or higher uncontrolled intercurrent illness

  * NOTE: To receive an agent, participant must not have any uncontrolled intercurrent illness requiring antibiotic/antiviral/antifungal therapy or interventional procedures. Participants with infections unlikely to be resolved within 2 weeks following registration should not be considered for the trial
* Participants must not have a known grade 2 or higher uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia
* Participants must not have any of the following:

  * Cirrhosis at a level of Child-Pugh B (or worse),
  * Cirrhosis (any degree) and a history of hepatic encephalopathy, or
  * Clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Participants must not be receiving any medications or substances that are inhibitors or inducers of CYP3A. Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug is prohibited.

  * NOTE: Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product. The participant wallet card should be presented to the participant
* Participants must not have baseline fasting glucose (after 8-hour fast) > 160 mg/dL (8.9 mmol/L) within 28 days prior to registration
* Participants with known diabetes mellitus must not require insulin therapy or have a baseline fasting glucose >150 mg/dL (8.3 mmol/L) or high glycosylated hemoglobin (Hb)A1c, (>= 8.0%), suggesting poorly controlled diabetes
* Participants who are on a stable dose of oral diabetes medication >= 2 weeks prior to initiation of study drug treatment are eligible for enrollment
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) must not have a potential to interfere with the safety or efficacy assessment of the investigational regimen
* Participants must not have lung disease requiring active systemic therapy or placing participants at increased risk of toxicity related to study-directed therapy including, but not limited to pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Participants must not be pregnant or nursing. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is of "reproductive potential". In addition to routine contraceptive methods, "effective contraception" also includes surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must not have psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  The proportion of participants who have a partial or complete response (confirmed or unconfirmed) as best response.

SECONDARY OUTCOMES:
Progression free survival | From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Response rates and associated confidence intervals will be calculated. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.
Overall survival | From date of registration to date of death due to any cause, assessed up to 3 years
  Response rates and associated confidence intervals will be calculated. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.
Duration of response | From date of first documentation of response (complete response, partial response, confirmed or unconfirmed) to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years
  Response rates and associated confidence intervals will be calculated. Will be estimated using the method of Kaplan-Meier. The Brookmeyer-Crowley method will be used to calculate confidence intervals for median times.

CONTACTS AND LOCATIONS:
Overall Officials: Reva K Basho, Principal Investigator — SWOG Cancer Research Network
Locations (210):
- United States (208):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - PCR Oncology, Arroyo Grande, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Saint John's Cancer Institute, Santa Monica, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Memorial Hospital, Marysville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - OhioHealth Westerville Medical Campus/Westerville Cancer Center, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Puerto Rico (2):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Centro Comprensivo de Cancer de UPR, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm